CLINICAL TRIAL: NCT01984645
Title: Identifying Primary Care Providers and Notifying Them Upon Admission of Their Patients to New York-Presbyterian Hospital
Brief Title: Primary-care-provider Identification And Notification
Acronym: PIANO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, David Vawdrey, Assistant Professor of Biomedical Informatics, Columbia University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAK1805
Record Dates: First submitted 2013-10-30; First posted 2013-11-15 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Emergency
Keywords: Emergency Visit; Secure Health messaging; Inpatient
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Notification (Experimental): Providers in this arm will receive a secure online notification whenever their patients are visited in the emergency department or admitted as an inpatient.
  Interventions: Other: Notification
- No intervention (No Intervention): Providers in this arm will not get a secure online notification about their patient's visit to the emergency department or inpatient admission.

INTERVENTIONS:
Other: Notification — Providers in the intervention group will receive a secure electronic notification when their patients are visited in the emergency department or admitted as an inpatient.
  Arms: Notification

SUMMARY:
New York-Presbyterian Hospital has created a system that notifies its primary care providers whenever their patients are admitted to the hospital. In this study, the investigators want to evaluate how accurate this system is and how it is affecting the primary providers and their health care delivery.

DETAILED DESCRIPTION:
The investigators will interview the participating providers to understand if they were aware of the admission of their patients, and how they want to get involved in the care of that patient while he/she is in hospital. The investigators will also look at the data in the Electronic Health Record system to understand how providers are acting in response to the notifications.

Lastly, the investigators will determine if the notifications have resulted in any change in the care of the patients, specifically in terms of the number of days from discharge until the next clinic visit.

ELIGIBILITY:
Inclusion Criteria:

* Primary Care Provider at the New York Presbyterian.

Exclusion Criteria:

* No clinic rotation during the study period

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7023 (Actual)
Dates: Start 2012-09; Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Mean duration until first post-discharge outpatient visit | 1 year
  The investigators will measure the time from each patient's discharge until their first follow-up visit in the outpatient setting. The investigators hypothesize that the automated notification will result is earlier post-discharge followups.

SECONDARY OUTCOMES:
Mean number of secure health messages (SHMs) | 1-7 days after each admission
  Once a primary care provider is notified about their patient's admission via a secure health message (SHM), the investigators will measure number of such SHMs that are read within 24 hours and within 7 days

OTHER OUTCOMES:
Average rate of readmission to inpatient setting | 1 year
  The investigators will compare the rate of readmission for patients associated with providers in the two arms of the study, to assess if provider's notification about their patient's visit to the emergency department has any effect on rate of readmission.

CONTACTS AND LOCATIONS:
Overall Officials: David K Vawdrey, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No